CLINICAL TRIAL: NCT00112424
Title: Clinical Trial of Cardiac Magnetic Resonance Imaging in Routine Evaluation Prior to Superior Cavo-Pulmonary Anastomosis
Brief Title: Trial of Cardiac Magnetic Resonance Imaging (MRI) Versus Cardiac Catheterization Prior to Glenn Operation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: David W. Brown, MD. Principal Investigator, Childrens Hospital Boston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CH 02-12-155
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Last update posted 2008-01-31 (Estimated); Status verified 2008-01

CONDITIONS: Congenital Heart Defects
Keywords: Superior cavo-pulmonary anastomosis; Glenn operation; Congenital heart defects; Cardiac magnetic resonance imaging
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Cardiac Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Diagnostic cardiac MRI — Routine cardiac MRI done under general anesthesia as pre-operative evaluation.
  Other Names: Cardiac Magnetic Resonance
Procedure: Cardiac catheterization — Routine cardiac catheterization prior to Glenn operation.
  Other Names: Cardiac cath.

SUMMARY:
This study is a prospective, randomized study of patients with single ventricle heart disease who are to undergo superior cavo-pulmonary anastomosis, or "Glenn" operation. Such patients have historically undergone cardiac catheterization to ensure suitability for the procedure. Cardiac magnetic resonance imaging (cardiac MRI) is a newer technology that provides excellent anatomic and functional imaging of the heart. This study is designed to demonstrate our hypothesis that cardiac magnetic resonance imaging will provide comparable information to catheterization, with less side effects.

DETAILED DESCRIPTION:
This is a prospective, randomized study of patients with single ventricle congenital heart disease presenting for superior cavo-pulmonary anastomosis, or "Glenn" operation. Such patients in the past have routinely undergone pre-operative invasive cardiac catheterization to assess anatomic and hemodynamic suitability for this procedure. Recent retrospective reviews, including our own (J Thorac Cardiovasc Surg 2003: July;126(1):272-81) have suggested that such catheterization may not benefit many patients, and that non-invasive assessment may allow adequate evaluation while avoiding many (typically minor) complications seen with cardiac catheterization in this high risk group of infants. Cardiac MRI is a non-invasive imaging modality that can deliver superior anatomic information (such as vascular and intracardiac anatomy) as well as functional data (ventricular volumes and ejection fraction), and may be a safe alternative to catheterization in such patients. In this study, patients undergo screening echocardiogram prior to enrollment in the study to assess degree of risk for the operation (such as pulmonary vein obstruction, a clear risk factor for poor outcome) or for demonstrated need for catheterization intervention (such as aortic arch obstruction requiring balloon dilation); patients with low risk echocardiograms whose parents grant informed consent for the study are then randomized in a prospective fashion to cardiac MRI or cardiac catheterization. The findings of each study are then reviewed by the subject's cardiologist and cardiac surgeon; patients in whom further pre-operative information may cross over to another study if deemed necessary (such as catheterization in patients in whom an unsuspected finding is noted, or cardiac MRI in patients in whom further functional data may be desired). Patients are followed for details of the hospital stay (including hospital length of stay, complications, hospital charges) for the pre-operative testing, as well as operative and post-operative outcomes (new/missed diagnoses, hospital stay, operative and post-operative complications, achievement of a clinical definition of a "good" outcome from the Glenn operation).

ELIGIBILITY:
Inclusion Criteria:

* Single ventricle heart disease patients presenting for Glenn operation

Exclusion Criteria:

* Aortic arch obstruction
* Pulmonary vein stenoses
* Severe ventricular dysfunction
* Pulmonary hypertension

Ages: 6 Weeks to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2004-01; Primary Completion 2006-06 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Toxicity profile for each group | 3 Months Post-Glenn operation

SECONDARY OUTCOMES:
Operative and post-operative outcomes | 30 days post-operation
Missed diagnoses | 3 months post-Glenn operation
Cost | Pre-operative evaluation
Clinical Definition of successful Glenn operation | 3 months post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: David W. Brown, MD, Principal Investigator — Childrens Hospital Boston
Locations (1):
- Childrens Hospital, Boston, Boston, Massachusetts, United States

REFERENCES:
- [Background] Brown DW, Gauvreau K, Moran AM, Jenkins KJ, Perry SB, del Nido PJ, Colan SD. Clinical outcomes and utility of cardiac catheterization prior to superior cavopulmonary anastomosis. J Thorac Cardiovasc Surg. 2003 Jul;126(1):272-81. doi: 10.1016/s0022-5223(03)00054-0. PMID 12878965
- [Background] Ro PS, Rychik J, Cohen MS, Mahle WT, Rome JJ. Diagnostic assessment before Fontan operation in patients with bidirectional cavopulmonary anastomosis: are noninvasive methods sufficient? J Am Coll Cardiol. 2004 Jul 7;44(1):184-7. doi: 10.1016/j.jacc.2004.02.058. PMID 15234431